CLINICAL TRIAL: NCT03021655
Title: Effectiveness of Using Adventure-based Training and WhatsApp Group to Relieve Emotion and Pressure so as to Quit Smoking: A Pilot Randomized Control Trial
Brief Title: A Pilot Randomized Control Trial to Help Youth Smokers to Quit Smoking:
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. LI William Ho Cheung, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: YouthQuitline_RCT
Record Dates: First submitted 2017-01-12; First posted 2017-01-16 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Smoking Cessation
Keywords: Youth; Randomized controlled trial; Adventure-based training; WhatsApp
MeSH Terms: conditions — Smoking Cessation | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Adventure-based intervention group (Experimental): Adventure-based intervention group included 1 day-camp and will be divided into 2 parts: (1) physical activity such as wall climbing, ropes course etc, (2) health education delivering about the relationship of self-efficacy, self-esteem, emotion and smoking abstinence. The training will be held before the 6-month follow-up. Telephone follow-up will be conducted at 1-week, 1-, 3-, 6-, 9-, 12- and 24-month.
  Interventions: Behavioral: Adventure-based intervention group
- WhatsApp intervention group (Experimental): For WhatsApp intervention group, not more than 8 subjects with same gender will be assigned into a group. Messages about mood and stress management will be sent to the group per week and the group will last for 6 months. It aims to relieve their pressure and emotion by sharing their unhappy things with other subjects. Telephone follow-up will be conducted at 1-week, 1-, 3-, 6-, 9-, 12- and 24-month.
  Interventions: Behavioral: WhatsApp intervention group
- Control group (Other): For the control group, the subjects will receive telephone counseling on quitting smoking at 1-week, 1-, 3-, 6-, 9-, 12- and 24-month.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Adventure-based intervention group — One-day adventure-based training will be assigned to subjects and the activities include wall climbing, rope course and health talk on mood, pressure management and smoking cessation.
  Arms: Adventure-based intervention group
Behavioral: WhatsApp intervention group — A WhatsApp group will be opened for the subjects and we will send messages about mood and pressure management to them and encourage them to quit smoking. The subjects can share their unhappy things in the group.
  Arms: WhatsApp intervention group
Behavioral: Control group — Telephone follow-up will be conducted at 1-week, 1-, 3-, 6-, 9-, 12-, 24-month and smoking cessation counselling will be delivered to the subjects.
  Arms: Control group

SUMMARY:
This study is a 3-arm randomized controlled trial including: (1) Adventure-based training intervention group, (2) WhatsApp intervention group and (3) Control group.

DETAILED DESCRIPTION:
Depression and stress are obstacles of youth smokers to quit smoking, youth smokers who have positive thinking and less depression exhibited smoking abstinence at last. Adventure-based training could enhance participants' self-efficacy, self-esteem and also improve mental health of children and youth by doing physical activity. On the other hand, previous mobile phone-based studies (e.g. short messaging services or Apps) showed that the mental health of youth had been improved by providing instant response to the subjects when they felt depressed. A paper published recently proved that WhatsApp group could prevent relapse among the quitters. Thus, adventure-based training and social support in WhatsApp group would predict to reduce depression and stress so as to quit smoking in youth.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong resident aged 25 or below
* Able to communicate, read and write in Cantonese/ Chinese
* Smoked in the past 30 days
* Mobile can access internet
* Would access internet through mobile or at home

Exclusion Criteria:

* Have difficulty to communicate via telephone
* Ever used/using psychiatric drugs
* Physically disabled
* Having queries irrelevant to tobacco control
* Undergoing other smoking cessation service

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-12; Primary Completion 2021-11 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Self-reported 7-day point prevalence | 6-month
  The subjects will be asked whether they have smoked cigarette in the past 7 day at 6-month

SECONDARY OUTCOMES:
Biochemical validated quit rate | 6-month
  Bio-chemical validated quit rate will be conducted if the subjects who reported they have been stop smoking for at least 7 days at 6-month. They will be invited to perform saliva cotinine test (using NicAlert strip) plus exhaled carbon monoxide text to validate the smoking status.
Change in Depressive symptoms | 6-month
  A 20-item scale (CESDC) will be used to assess the depressive symptoms of the subjects after 6 months.
Change in Self-esteem | 6-month
  A 10-item scale (RSES) will be used to assess the self-esteem level of the subjects after 6 months.
Change in Quality of life | 6-month
  A 11-item scale (SF-6D) will be used to assess the quality of life of the subjects after 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ho-cheung Li, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No